CLINICAL TRIAL: NCT06032468
Title: ARC Intellicare for Telerehabilitation in Neurological Patients
Brief Title: ARC Intellicare for Telerehabilitation
Acronym: ARCTRAN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5135
Record Dates: First submitted 2023-05-12; First posted 2023-09-13 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2023-05

CONDITIONS: Parkinson Disease; Multiple Sclerosis; Stroke
MeSH Terms: conditions — Parkinson Disease; Multiple Sclerosis; Stroke

STUDY DESIGN:
Intervention Model Description: Early feasibility study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rehabilitation with ARC Intellicare Device (Experimental): rehabilitation exercise for 8 weeks using wearable devices
  Interventions: Device: ARC Intellicare
- Rehabilitation with exercise sheet (Active Comparator): rehabilitation exercise for 8 weeks using rehabilitation exercise sheets
  Interventions: Other: Rehabilitation sheets

INTERVENTIONS:
Device: ARC Intellicare — wearable devices to guide rehabilitation exercise
  Arms: Rehabilitation with ARC Intellicare Device
Other: Rehabilitation sheets — rehabilitation exercise sheets to guide rehabilitation exercise
  Arms: Rehabilitation with exercise sheet

SUMMARY:
In the last 5 years, the available literature evidence has indicated that, in terms of clinical efficacy, telerehabilitation can give comparable results compared to face-to-face rehabilitation. Studies of post-stroke patients have revealed some benefits of telerehabilitation, such as the ability for patients to self-record pain, mood and activity. Telerehabilitation has comparable efficacy to face-to-face rehabilitation for the recovery of some abilities, such as motor function, Activities of Daily Living (ADL), and independence; it is less effective, however, for the recovery of balance control. Published reviews concerning, in particular, neurological/neurodegenerative diseases show that telerehabilitation systems are effective in maintaining and/or improving some motor aspects, such as balance and gait, and non-motor aspects, such as mood and quality of life; they also increase patient satisfaction, so in the long term they appear to be beneficial, convenient and satisfying for patients and operators.

ARC Intellicare is a device undergoing certification as a Class I Medical Device (DM), already clinically tested during two uncontrolled clinical feasibility studies: ARCANGEL study (post-stroke, ClinicalTrials.gov Identifier: NCT03787433) and RICOMINCIARE study (post-COVID19 and Parkinson's disease, ClinicalTrials.gov Identifier: NCT05074771).

ELIGIBILITY:
Inclusion Criteria:

* patients with diagnosis of Parkinson's disease with Hoehn&Yahr staging 1-3
* diagnosis of multiple sclerosis with extended disability scale score 3.5-6
* diagnosis of ischemic stroke in the past 12 months

Exclusion Criteria:

* history of falls
* dementia
* epilepsy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2023-01-09 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Efficacy outcome: Six minutes walking test (6MWT) | 8 weeks
  number of meters walked in brisk 6 minutes walk
Efficacy outcome: Borg scale | 8 weeks
  score 0-20 of perceived effort during a motor task (higher scores mean a better or worse outcome)
safety outcome: adverse event frequency | 8 weeks
  number of adverse events reported
Usability outcome: adherence to prescription | 8 weeks
  percent of rehabilitation sessions completed

CONTACTS AND LOCATIONS:
Locations (1):
- policlinico Universitario A Gemelli, Roma, Rome, Italy

IPD SHARING:
Plan to Share IPD: No